CLINICAL TRIAL: NCT01613040
Title: A Multiple-center, Multiple-dose, Randomized, Double-blind, Double-dummy, Placebo-controlled, Positive-controlled, Parallel Group Study to Investigate the Effect of RO4917838 on the QTc Interval in Healthy Subjects.
Brief Title: A Study of the Effect of RO4917838 on the QTcF Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP21705; 2008-001127-57 (EudraCT Number)
Record Dates: First submitted 2012-05-23; First posted 2012-06-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: RO4917838
- Treatment B (Experimental)
  Interventions: Drug: RO4917838
- Treatment C (Placebo Comparator)
  Interventions: Drug: Moxifloxacin; Drug: RO4917838 placebo
- Treatment D (Placebo Comparator)
  Interventions: Drug: Moxifloxacin; Drug: RO4917838 placebo

INTERVENTIONS:
Drug: Moxifloxacin — Single oral dose on Day 1
  Arms: Treatment C
Drug: Moxifloxacin — Single oral dose on Day 11
  Arms: Treatment D
Drug: RO4917838 — Multiple daily low doses of RO4917838 for 10 days
  Arms: Treatment A
Drug: RO4917838 — Multiple daily oral high doses of RO4917838 for 10 days
  Arms: Treatment B
Drug: RO4917838 placebo — Oral daily doses of placebo to RO4917838 for 10 days
  Arms: Treatment C; Treatment D

SUMMARY:
This multiple-center, multiple-dose, randomized, double-blind, double-dummy, placebo-controlled, positive-controlled, parallel group study will investigate the effect of RO4917838 on the QTc interval in healthy volunteers. Healthy volunteers will be randomized to one of 4 treatment arms; Arm A: low dose of RO4917838, Arm B: high dose of RO4917838, Arm C: placebo to RO4917838 and moxifloxacin on Day 1, Arm D: placebo to RO4917838 and moxifloxacin on Day 11. The anticipated time on study treatment is 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 65 years inclusive
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive.
* Have no contraindications from the following: a detailed medical and surgical history, and a complete physical examination
* Able to participate, and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, mental, cardiac, vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis.
* History of alcohol and/or drug abuse or addiction within the last 2 years prior to Day 1 of the study.
* Consumption of nicotine and/or tobacco containing products within the last 3 months prior to Day 1 of the study.
* Infection with human immunodeficiency virus, hepatitis B and/or hepatitis C
* Any condition or disease detected during the medical interview / physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator.
* Positive drug screen or alcohol test at screening or prior to enrollment.
* Coffee or tea consumption > 10 cups per day or methylxanthine containing drinks >1.5 liter/day or more than 250 g/day of chocolate.
* Alcohol consumption averaging > 3 drinks daily

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes in QTcF interval at steady state | Baseline and Day 10

SECONDARY OUTCOMES:
Change of electrocardiogram | Baseline and Day 10
Correlation of RO4917838 plasma concentration and the electrocardiogram | Day 10
Change in the QTc interval, using moxifloxacin as an active control | Days 1 and 11
Safety: incidence of adverse events | 8 weeks
Pharmacokinetics: area under the concentration time curve of RO4917838 | Up to Day 19
Pharmacokinetics: Maximum plasma concentration of RO4917838 | Up to Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Tempe, Arizona, United States
- Strasbourg, France

REFERENCES:
- [Derived] Hofmann C, Banken L, Hahn M, Swearingen D, Nagel S, Martin-Facklam M. Evaluation of the effects of bitopertin (RG1678) on cardiac repolarization: a thorough corrected QT study in healthy male volunteers. Clin Ther. 2012 Oct;34(10):2061-71. doi: 10.1016/j.clinthera.2012.08.010. Epub 2012 Sep 12. PMID 22980315